CLINICAL TRIAL: NCT04934267
Title: The Effect of Joint Hypermobility Syndrome on Delayed Onset of Muscle Soreness and Recovery Time
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: New York Institute of Technology (Other)
Responsible Party: Principal Investigator, Peter Douris, Professor, New York Institute of Technology
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: BHS-1636
Record Dates: First submitted 2021-05-19; First posted 2021-06-22 (Actual); Last update posted 2021-11-02 (Actual); Status verified 2021-11

CONDITIONS: Hypermobility Syndrome
Keywords: DOMS; Hypermobility,; Recovery

STUDY DESIGN:
Intervention Model Description: Comparing the recovery times and length of DOMS in individuals with JHS to individuals with normal ranges of motion in response to exercise
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Eccentric exercise of elbow in order to induce Delayed Onset of Muscle Soreness (Experimental): There will be two groups, an experimental group with hypermobile individuals, and a control group with individuals that are not hypermobile with normal ranges of motion. All participants will take part in an exercise session with eccentric bicep curls based on their 1 repetition maximum (1RM).Both groups will perform 1 set of standing eccentric bicep curls based on their 1RM to failure in order to induce DOMS.The exercise will stop when the participant cannot volitionally keep up with the 5 second count lowering the weight. Prior to exercise, baseline measurements will be taken for all dependent variables. These measures will be taken every day at the same time of day,for the next 4 days.
  Interventions: Other: Eccentric Exercise for subjects with JHS; Other: Eccentric Exercise for Controls

INTERVENTIONS:
Other: Eccentric Exercise for subjects with JHS — There will be two groups, an experimental group with hypermobile individuals, and a control group with individuals that are not hypermobile with normal ranges of motion. All participants will take part in an exercise session with eccentric bicep curls based on their 1 repetition maximum (1-RM), which is the highest amount of weight that they can lift concentrically once. The independent variables are the two groups and the dependent variables are girth, resting arm angle, Pain, McGill Pain Questionnaire, and pressure pain threshold. This groups will perform 1 set of standing eccentric bicep curls order to induce DOMS.Each rep will include a timed 5 second long eccentric component without an concentric component,. The exercise will stop when the participant cannot volitionally keep up with the 5 second count. Prior to exercise, baseline measurements will be taken for all dependent variables. These measures will be taken every day at the same time of day,for the next 4 days.
Other: Eccentric Exercise for Controls — There will be two groups, an experimental group with hypermobile individuals, and a control group with individuals that are not hypermobile with normal ranges of motion. All participants will take part in an exercise session with eccentric bicep curls based on their 1 repetition maximum (1-RM), which is the highest amount of weight that they can lift concentrically once. The independent variables are the two groups and the dependent variables are girth, resting arm angle, Pain, McGill Pain Questionnaire, and pressure pain threshold. This groups will perform 1 set of standing eccentric bicep curls order to induce DOMS.Each rep will include a timed 5 second long eccentric component without an concentric component,. The exercise will stop when the participant cannot volitionally keep up with the 5 second count. Prior to exercise, baseline measurements will be taken for all dependent variables. These measures will be taken every day at the same time of day,for the next 4 days.

SUMMARY:
The purpose of the study is to investigate Joint Hypermobility Syndrome (JHS) and its effect on delayed onset muscle soreness (DOMS) and recovery time. The hypothesis is that people with JHS will experience increased DOMS when compared to non-hypermobile people. The results this study may assist and add to the body of knowledge when treating and exercising patients with JHS, as considerations can possibly be made when treating this population. Subjects with JHS may experience greater DOMS and require more time to recover between treatment sessions.

DETAILED DESCRIPTION:
The research design will be a 2x5 factorial design. There will be two groups, an experimental group with hypermobile individuals, and a control group with individuals that are not hypermobile with normal ranges of motion. All participants will take part in an exercise session with eccentric bicep curls based on their 1 repetition maximum (1-RM), which is the highest amount of weight that they can lift concentrically once. The independent variables are the two groups and the dependent variables are girth, resting arm angle (RANG), Pain 1-10 Visual Analogue Scale (VAS), McGill Pain Questionnaire, and pressure pain threshold using an algometer. The proposed study will include 20 participants between the ages of 18-35 years old, who exercise recreationally. Both groups will perform 1 set of standing eccentric bicep curls based on their 1RM to failure in order to induce DOMS.7 Each rep will include a timed 5 second long eccentric component with a metronome and without an concentric component, as the research conductors will lift the weight up or concentrically for the participant. The exercise will stop when the participant cannot volitionally keep up with the 5 second count lowering the weight. Prior to exercise, baseline measurements will be taken for all dependent variables. These measures will be taken every day at the same time of day,for the next 4 days. Girth is the measurement of the circumference of a limb measuring swelling, which commonly occurs during DOMS.7 Resting Arm Angle (RANG) is a range of motion (ROM) measurement of the arm while resting.The VAS is a simple pain scale ranging from 0-10, 0 being no pain and 10 being the worst pain the participant has felt..The McGill Pain Questionnaire is a questionnaire that allows the participant to rate their pain'.7 Lastly, the pressure pain threshold using an algometer is done by applying continuous ascending pressure at a constant rate in order to quantify the individuals pain pressure threshold.The change in measurements from baseline to post exercise will be recorded for subsequent data analysis.

ELIGIBILITY:
Inclusion Criteria:

1. Age range: 18-35 years
2. Good overall health
3. Regularly participate in recreational exercise
4. 10 subjects with normal ranges of motion (score of <4 on Beighton Scale), 10 subjects with increased ranges of motion (score of >4 on Beighton Scale AND hypermobile in the elbow)

Exclusion Criteria:

1. Individuals with Ehler-Danlos Syndrome.
2. Any major musculoskeletal injuries in the last 6 months.
3. Any recent traumas that could lead to acute hypermobility or instabilities
4. Any known disorders that impede recovery/healing time (i.e. Lupus, Rheumatoid Arthritis, Scleroderma).
5. Any other health issues that would risk the safety of the subject.

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Estimated)
Dates: Start 2021-05-01 (Actual); Primary Completion 2022-05-01 (Estimated); Study Completion 2022-05-15 (Estimated)

PRIMARY OUTCOMES:
"Change" is being assessed in Girth between the 5 time points | Baseline (Day 1) through Day 2,3,4 and 5.
  Girth is the measurement of the circumference of a limb in centimetres, measuring edema, which commonly occurs during DOMS.
"Change' is being assessed in Resting arm angle (RANG)between the 5 time points, | Baseline (Day 1) through Day 2,3,4 and 5.
  Resting Arm Angle (RANG) is a Range Of Motion measurement in degrees of the arm while resting
"Change" is being assessed in Visual Analogue Scale (VAS) of Pain between the 5 time points | Baseline (Day 1) through Day 2,3,4 and 5.
  The VAS is a simple pain scale ranging from 0-100 mm, 0 being no pain and 100 mm being the worst pain the participant has felt.
"Change" is being assessed in The McGill Pain Questionnaire (SF-MQ2)between the 5 time points | Baseline (Day 1) through Day 2,3,4 and 5.
  The McGill Pain Questionnaire (SF-MQ2) is a questionnaire that allows the participant to rate their pain.
"Change" is being assessed in Algometer pain pressure threshold between the 5 time points | Baseline (Day 1) through Day 2,3,4 and 5.
  the pressure pain threshold using an algometer is done by applying continuous ascending pressure at a constant rate on their self reported most painful area surrounding the elbow in order to quantify the individuals pain pressure threshold, measured in kg.

CONTACTS AND LOCATIONS:
Overall Officials: Peter C Douris, EdD, Principal Investigator — New York Institute of Technology
Locations (1):
- New York Institute of Technology, Old Westbury, New York, United States

IPD SHARING:
Plan to Share IPD: No
No plan

REFERENCES:
- [Background] Tinkle BT, Levy HP. Symptomatic Joint Hypermobility: The Hypermobile Type of Ehlers-Danlos Syndrome and the Hypermobility Spectrum Disorders. Med Clin North Am. 2019 Nov;103(6):1021-1033. doi: 10.1016/j.mcna.2019.08.002. PMID 31582002
- [Background] Lee H, Petrofsky JS, Laymon M, Yim J. A greater reduction of anterior cruciate ligament elasticity in women compared to men as a result of delayed onset muscle soreness. Tohoku J Exp Med. 2013 Oct;231(2):111-5. doi: 10.1620/tjem.231.111. PMID 24107654
- [Background] Castori M, Morlino S, Celletti C, Celli M, Morrone A, Colombi M, Camerota F, Grammatico P. Management of pain and fatigue in the joint hypermobility syndrome (a.k.a. Ehlers-Danlos syndrome, hypermobility type): principles and proposal for a multidisciplinary approach. Am J Med Genet A. 2012 Aug;158A(8):2055-70. doi: 10.1002/ajmg.a.35483. Epub 2012 Jul 11. PMID 22786715
- [Background] Terry RH, Palmer ST, Rimes KA, Clark CJ, Simmonds JV, Horwood JP. Living with joint hypermobility syndrome: patient experiences of diagnosis, referral and self-care. Fam Pract. 2015 Jun;32(3):354-8. doi: 10.1093/fampra/cmv026. Epub 2015 Apr 24. PMID 25911504
- [Background] Douris P, Southard V, Ferrigi R, Grauer J, Katz D, Nascimento C, Podbielski P. Effect of phototherapy on delayed onset muscle soreness. Photomed Laser Surg. 2006 Jun;24(3):377-82. doi: 10.1089/pho.2006.24.377. PMID 16875447